CLINICAL TRIAL: NCT02755597
Title: A Phase 3, Multicenter, Randomized, Double Blind Study of Bortezomib and Dexamethasone in Combination With Either Venetoclax or Placebo in Subjects With Relapsed or Refractory Multiple Myeloma Who Are Sensitive or Naïve to Proteasome Inhibitors
Brief Title: A Study Evaluating Venetoclax (ABT-199) in Multiple Myeloma Subjects Who Are Receiving Bortezomib and Dexamethasone as Standard Therapy
Acronym: Bellini
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-031; 2015-004411-20 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2016-04-20; First posted 2016-04-29 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Relapsed/refractory multiple myeloma; Relapsed multiple myeloma; Refractory multiple myeloma; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — venetoclax; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venetoclax + Bortezomib and Dexamethasone (Experimental): Cycles 1-8: Venetoclax 800 mg orally every day (QD) on Days 1 - 21 plus bortezomib 1.3 mg/m^2 subcutaneously or IV on Days 1, 4, 8 & 11 and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11 & 12; Cycles 9 and beyond: Venetoclax 800 mg orally every day (QD) on Days 1 - 35 plus bortezomib 1.3 mg/m^2 subcutaneously or IV on Days 1, 8, 15 and 22 and dexamethasone 20 mg orally on Days 1, 2, 8, 9, 15, 16, 22 and 23
  Interventions: Drug: Venetoclax; Drug: Bortezomib; Drug: Dexamethasone
- Placebo + Bortezomib and Dexamethasone (Placebo Comparator): Cycles 1-8: Placebo (to match venetoclax 100 mg tablet) 800 mg orally every day (QD) on Days 1 - 21 plus bortezomib 1.3 mg/m^2 subcutaneously or IV on Days 1, 4, 8 & 11 and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11 & 12; Cycles 9 and beyond: Placebo (to match venetoclax 100 mg tablet) 800 mg orally every day (QD) on Days 1 - 35 plus bortezomib 1.3 mg/m^2 subcutaneously or IV on Days 1, 8, 15 and 22 and dexamethasone 20 mg orally on Days 1, 2, 8, 9, 15, 16, 22 & 23
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Placebo for venetoclax

INTERVENTIONS:
Drug: Venetoclax — Participants self-administered venetoclax tablets by mouth QD in combination with bortezomib. Venetoclax was to be given before other agents administered on the same day, if applicable. Each venetoclax dose was to be taken all at one time with approximately 240 mL of water within 30 minutes after completion of breakfast or the subject's first meal of the day. Tablets were to be swallowed whole and must not have been broken, chewed, or crushed. On days that pre-dose PK sampling was required, dosing occurred at the clinic to facilitate PK sampling.
  Other Names: VENCLEXTA; VENCLYXTO
  Arms: Venetoclax + Bortezomib and Dexamethasone
Drug: Bortezomib — Bortezomib (subcutaneous injection [preferred] or IV) was given following administration of venetoclax or placebo in Cycles 1 -8 on Days 1, 4, 8 and 11, and for Cycles 9 and beyond, on Days 1, 8, 15 and 22 and was to be administered per the prescribing information. The route of administration was to stay the same during the study.
  Other Names: Velcade
Drug: Dexamethasone — Dexamethasone was to be given orally, administered per the prescribing information, the day of bortezomib dosing and the following day, given the protocol-defined dosing window (bortezomib dosing window is ± 1 day) is maintained. If bortezomib was interrupted or a dose is skipped, dexamethasone was to be administered as scheduled per protocol (unless dexamethasone was interrupted due to toxicity).
Drug: Placebo for venetoclax — Participants self-administered placebo tablets by mouth QD in combination with bortezomib. Placebo was to be given before other agents administered on the same day, if applicable. Each placebo dose was to be taken all at one time with approximately 240 mL of water within 30 minutes after completion of breakfast or the subject's first meal of the day. Tablets were to be swallowed whole and must not have been broken, chewed, or crushed. On days that pre-dose PK sampling was required, dosing occurred at the clinic to facilitate PK sampling.
  Arms: Placebo + Bortezomib and Dexamethasone

SUMMARY:
This was a Phase 3, multicenter, randomized, double blind, placebo-controlled study evaluating the efficacy and safety of venetoclax plus bortezomib and dexamethasone in participants with relapsed or refractory multiple myeloma who are considered sensitive or naïve to proteasome inhibitors and received 1 to 3 prior lines of therapy for multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
* Participant has documented relapsed or progressive multiple myeloma on or after any regimen or who are refractory to the most recent line of therapy. Relapsed myeloma is defined as previously treated myeloma that progresses and requires initiation of salvage therapy, but does not meet the criteria for refractory myeloma. Refractory myeloma is defined as disease that is nonresponsive (failure to achieve minimal response or development of progressive disease [PD]) while on primary or salvage therapy, or progresses within 60 days of last therapy.
* Participant must have received prior treatment with at least one, but no more than three, prior lines of therapy for multiple myeloma. A line of therapy consists of ≥ 1 complete cycle of a single agent, a regimen consisting of combination of several drugs, or a planned sequential therapy of various regimens.
* Prior treatment with bortezomib or other proteasome inhibitor is allowed, provided ALL of the following criteria are met: Disease is NOT refractory to any proteasome inhibitor, defined as no disease progression (i.e., PD, per International Myeloma Working Group [IMWG] or European Society for Blood and Marrow Transplantation [EBMT] criteria) while receiving proteasome inhibitor therapy or within 60 days after the last dose, AND best response achieved with any proteasome inhibitor therapy (alone or in combination) was at least a Partial Response (PR), AND participant did not discontinue any proteasome inhibitor due to intolerance or ≥ Grade 3 related toxicity.
* Participant has measurable disease at Screening, defined as at least one of the following: Serum M-protein ≥ 0.5 g/dL, OR Urine M-protein ≥ 200 mg in 24-hours, OR serum immunoglobulin free light chain (FLC) ≥ 10 mg/dL provided serum FLC ratio is abnormal.

Exclusion Criteria:

* Participant is refractory to any proteasome inhibitor, defined as progression on or within 60 days of the last dose of a proteasome inhibitor-containing regimen.
* Participant has had prior treatment with proteasome inhibitor within 60 days prior to first dose of study drug.
* Participant has any of the following conditions:

Non-secretory multiple myeloma, active plasma cell leukemia i.e., either 20% of peripheral white blood cells or greater than 2.0 X 10^9/liter (L) circulating plasma cells by standard differential, Waldenstrom's macroglobulinemia, amyloidosis, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), known Human Immunodeficiency Viral (HIV) infection, active hepatitis B or C infection based on blood screen tests, significant cardiovascular disease, including uncontrolled angina, severe or uncontrolled arrhythmia, recent myocardial infarction within 6 months of randomization, or congestive heart failure New York Heart Association (NYHA) Class ≥ 3, major surgery within 4 weeks prior to randomization, acute infections requiring parenteral therapy (antibiotic, antifungal, or antiviral) within 14 days prior to randomization, peripheral neuropathy ≥ Grade 3 or ≥ Grade 2 with pain within 2 weeks prior to randomization, uncontrolled diabetes or uncontrolled hypertension within 14 days prior to randomization, any other medical condition that, in the opinion of the Investigator, would adversely affect the participant's participation in the study

* Participant has a history of other active malignancies, including myelodysplastic syndrome (MDS), within the past 3 years prior to study entry, with the following exceptions: Adequately treated in situ carcinoma of the cervix uteri or the breast, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, prostate cancer Gleason grade 6 or lower AND with stable Prostate Specific Antigen (PSA) levels off treatment, previous malignancy with no evidence of disease confined and surgically resected (or treated with other modalities) with curative intent and unlikely to impact survival during the duration of the study
* If participant had prior allogeneic stem cell transplant (SCT), participant has evidence of ongoing graft-versus-host disease (GvHD)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (97):
- United States (4):
  - Rocky Mountain Regional VA Medical Center/Eastern Colorado Health Care System /ID# 156524, Aurora, Colorado
  - Univ of Colorado Cancer Center /ID# 149130, Aurora, Colorado
  - Duke Cancer Center /ID# 149099, Durham, North Carolina
  - Gabrail Cancer Center Research /ID# 149098, Canton, Ohio
- Australia (11):
  - Royal Prince Alfred Hospital /ID# 149108, Camperdown, New South Wales
  - Concord Repatriation General Hospital /ID# 149106, Concord, New South Wales
  - Liverpool Hospital /ID# 149110, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 149105, Herston, Queensland
  - The Queen Elizabeth Hospital /ID# 149104, Woodville South, South Australia
  - Royal Hobart Hospital /ID# 149111, Hobart, Tasmania
  - Box Hill Hospital /ID# 149112, Box Hill, Victoria
  - Peter MacCallum Cancer Ctr /ID# 149107, Melbourne, Victoria
  - Alfred Health /ID# 150085, Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 148967, Murdoch, Western Australia
  - Perth Blood Institute Ltd /ID# 148966, Nedlands, Western Australia
- Brazil (6):
  - Hospital das Clinicas da Universidade Federal de Goiás /ID# 149290, Goiânia, Goiás
  - Liga Norte Riograndense Contra o Câncer /ID# 149023, Natal, Rio Grande do Norte
  - Hospital Sao Lucas da PUCRS /ID# 149027, Porto Alegre, Rio Grande do Sul
  - Clinica Sao Germano /ID# 149851, São Paulo, São Paulo
  - Instituto Nacional de Câncer José Alencar Gomes da Silva (INCA) /ID# 149020, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo /ID# 149025, São Paulo
- Canada (2):
  - Victoria Hospital /ID# 149846, London, Ontario
  - CISSS de la Monteregie /ID# 149844, Greenfield Park, Quebec
- France (5):
  - CHU Limoges - Dupuytren 1 /ID# 149292, Limoges, Franche-Comte
  - CHU de Nantes, Hotel Dieu -HME /ID# 149294, Nantes, Pays de la Loire Region
  - Duplicate_Centre Hospitalier Lyon Sud /ID# 149300, Pierre-Bénite, Rhone
  - CHRU de Brest - Hopital Morvan /ID# 149299, Brest
  - CHU Grenoble - Hopital Michallon /ID# 149301, La Tronche
- Germany (3):
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 148949, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 148948, Dresden
  - Asklepios Klinik Altona /ID# 150116, Hamburg
- Hungary (5):
  - Debreceni Egyetem Klinikai Kozpont /ID# 152517, Debrecen, Hajdú-Bihar
  - Somogy Megyei Kaposi Mor Oktato Korhaz /ID# 152516, Kaposvár, Somogy County
  - Semmelweis Egyetem /ID# 152519, Budapest
  - Semmelweis Egyetem /ID# 152520, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 152518, Budapest
- University Hospital Galway /ID# 149061, Galway, Ireland
- Italy (5):
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 148939, Rome, Lazio
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 148942, Ancona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 148936, Bologna
  - Ospedale S.Eugenio /ID# 148938, Rome
  - A.O.U. Città della Salute e della Scienza di Torino/Ospedale Molinette /ID# 148943, Turin
- Japan (19):
  - Nagoya City University Hospital /ID# 150943, Nagoya, Aichi-ken
  - Kyushu University Hospital /ID# 150896, Fukuoka, Fukuoka
  - Ogaki Municipal Hospital /ID# 150783, Ogaki-shi, Gifu
  - Gunma University Hospital /ID# 150275, Maebashi, Gunma
  - National Hospital Organization Shibukawa Medical Center /ID# 150281, Shibukawa-shi, Gunma
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 150242, Hiroshima, Hiroshima
  - Kobe City Medical Center General Hospital /ID# 150944, Kobe, Hyōgo
  - National Hospital Organization Mito Medical Center /ID# 151051, Higashi Ibaraki-gun, Ibaraki
  - Duplicate_Kyoto Prefectural University of Medicine /ID# 150719, Kyoto, Kyoto
  - JCHO Kyoto Kuramaguchi Medical /ID# 150781, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 150945, Sendai, Miyagi
  - Okayama Medical Center /ID# 150717, Okayama, Okayama-ken
  - Japanese Red Cross Osaka Hospital /ID# 150716, Osaka, Osaka
  - Saitama Medical Center /ID# 151044, Kawagoe-shi, Saitama
  - Tochigi Cancer Center /ID# 150192, Utsunomiya, Tochigi
  - National Cancer Center Hospital /ID# 151039, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 150780, Koto-ku, Tokyo
  - Japanese Red Cross Medical Center /ID# 149902, Shibuya-ku, Tokyo
  - National Hospital Organization Disaster Medical Center /ID# 150784, Tachikawa-shi, Tokyo
- Russia (7):
  - Kuzbass Regional Clinical Hospital /ID# 148955, Kemerovo, Kemerovo Oblast
  - State Institution of Health of the Ryazan Regional Clinical Hospital /ID# 148956, Ryazan, Ryazan Oblast
  - LLC Novaya Klinika /ID# 148974, Pyatigorsk, Stavropol Kray
  - Central Clinical Hospital RZHD Medicine /ID# 148954, Moscow
  - Clinical Oncology Dispensary of Omsk /ID# 148953, Omsk
  - Samara State Medical University /ID# 148952, Samara
  - Bashkir State Medical University /ID# 151206, Ufa
- South Korea (8):
  - National Cancer Center /ID# 150889, Goyang, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 150888, Seongnam, Gyeonggido
  - Duplicate_Yonsei University Health System, Severance hospital. /ID# 150891, Seoul, Seoul Teugbyeolsi
  - Chonnam National University Hospital /ID# 150894, Gwangju
  - Gachon University Gil Medical Center /ID# 150893, Incheon
  - Seoul National University Hospital /ID# 150890, Seoul
  - Samsung Medical Center /ID# 150892, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital /ID# 150895, Seoul
- Spain (4):
  - Hospital Duran i Reynals /ID# 148989, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de la Princesa /ID# 148980, Madrid
  - Hospital Universitario 12 de Octubre /ID# 148981, Madrid
  - Hospital Universitario Dr. Peset /ID# 148986, Valencia
- Taiwan (4):
  - Changhua Christian Hospital /ID# 154447, Changhua City, Changhua County
  - China Medical University Hospital /ID# 154446, Taichung
  - National Taiwan University Hospital /ID# 154444, Taipei
  - Taipei Veterans General Hosp /ID# 154445, Taipei
- Ukraine (3):
  - Communal Nonprofit Enterprise Cherkasy Regional Oncology Dispensary /ID# 152414, Cherkasy
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council /ID# 152411, Dnipro
  - National Cancer Institute /ID# 152413, Kyiv
- United Kingdom (10):
  - Leicester Royal Infirmary /ID# 149057, Leicester, England
  - Barts Health NHS Trust /ID# 149050, London, London, City of
  - Nottingham University Hospitals NHS Trust /ID# 149047, Nottingham, Nottinghamshire
  - Blackpool Teaching Hospitals NHS Foundation Trust /ID# 149058, Blackpool
  - East Kent Hospitals University NHS Foundation Trust /ID# 149059, Canterbury
  - University College London Hospitals NHS Foundation Trust /ID# 149044, London
  - King's College Hospital NHS Foundation Trust /ID# 149045, London
  - Manchester University NHS Foundation Trust /ID# 149046, Manchester
  - Barking, Havering and Redbridge University Hospitals NHS Trust /ID# 149055, Romford
  - The Royal Wolverhampton NHS Trust /ID# 149043, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Kumar SK, Harrison SJ, Cavo M, de la Rubia J, Popat R, Gasparetto C, Hungria V, Salwender H, Suzuki K, Kim I, Onishi M, Ku G, Pothacamury R, Jalaluddin M, Zeng J, Ross JA, Dobkowska E, Moreau P. Venetoclax or placebo in combination with bortezomib and dexamethasone in relapsed or refractory multiple myeloma (BELLINI): final overall survival results from a randomised, phase 3 study. Lancet Haematol. 2025 Aug;12(8):e574-e587. doi: 10.1016/S2352-3026(25)00139-5. Epub 2025 Jun 27. PMID 40587991
- [Derived] Kumar SK, Harrison SJ, Cavo M, de la Rubia J, Popat R, Gasparetto C, Hungria V, Salwender H, Suzuki K, Kim I, Punnoose EA, Hong WJ, Freise KJ, Yang X, Sood A, Jalaluddin M, Ross JA, Ward JE, Maciag PC, Moreau P. Venetoclax or placebo in combination with bortezomib and dexamethasone in patients with relapsed or refractory multiple myeloma (BELLINI): a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1630-1642. doi: 10.1016/S1470-2045(20)30525-8. Epub 2020 Oct 29. PMID 33129376

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-To-Treat (ITT) analysis set: all randomized participants, analyzed by treatment group assignment given at the time of randomization
Period: Overall Study
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Started | 194 | 97
Completed | 0 | 0
Not Completed | 194 | 97
Not completed — Withdrew consent | 27 | 11
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 78 | 36
Not completed — Study terminated by Sponsor | 67 | 47
Not completed — Other, not specified | 20 | 3
Not completed — Participant missing reason for study discontinuation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) analysis set: all randomized participants, analyzed by treatment group assignment given at the time of randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone | Total
Number analyzed (Participants) | 194 | 97 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.41) | 65.9 (7.81) | 65.9 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 42 | 139
  Male | 97 | 55 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 7 | 32
  Not Hispanic or Latino | 169 | 90 | 259
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 28 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 124 | 66 | 190
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Time since diagnosis [Median (Full Range); unit: days] | 1263.5 [62.0 to 8356.0] | 1461.0 [195.0 to 4906.0] | 1318.0 [62.0 to 8356.0]
Number of prior lines of therapy [Median (Full Range); unit: number of prior lines of therapy] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
Number of prior lines of multiple myeloma therapy [Count of Participants; unit: Participants]
  1 line | 91 | 44 | 135
  2-3 lines | 103 | 53 | 156
Prior exposure to proteasome inhibitors (PI) [Count of Participants; unit: Participants]
  Refractory | 0 | 2 | 2
  Sensitive | 131 | 66 | 197
  Naïve | 61 | 28 | 89
  Unknown | 2 | 0 | 2
  MISSING | 0 | 1 | 1
Prior exposure to an immunomodulatory drug (IMID) [Count of Participants; unit: Participants]
  Refractory | 64 | 36 | 100
  Sensitive | 67 | 29 | 96
  Naïve | 63 | 30 | 93
  Unknown | 0 | 1 | 1
  MISSING | 0 | 1 | 1
Prior exposure to an anti-CD38 monoclonal antibody [Count of Participants; unit: Participants]
  Refractory | 5 | 1 | 6
  Sensitive | 0 | 0 | 0
  Naïve | 185 | 95 | 280
  Unknown | 0 | 0 | 0
  MISSING | 4 | 1 | 5
Multiple myeloma International Staging System(ISS) stage [Count of Participants; unit: Participants] — The International Staging System for multiple myeloma:
  Stage I: Serum β2 microglobulin (Sβ2M), < 3.5 mg/L; serum albumin ≥ 3.5 g/dL
  Stage II: Not ISS Stage I or III
  Stage III: Sβ2M > 5.5 mg/L
  Stage I represents the mildest form of multiple myeloma (best prognosis) and Stage III the most severe form (worst prognosis).
  Participants
    Stage I | 81 | 48 | 129
    Stage II | 69 | 32 | 101
    Stage III | 39 | 13 | 52
    Not evaluable | 5 | 3 | 8
    MISSING | 0 | 1 | 1
Chromosomal abnormality (CA) risk by fluorescent in situ hybridization (FISH) [Count of Participants; unit: Participants] — A 4 mL bone marrow aspirate sample was collected for baseline assessment of chromosomal abnormalities, including t(11;14), t(4;14), t(14;16), del 17p, 5+, 9+, 15+
  Participants
    High | 31 | 18 | 49
    Standard | 141 | 72 | 213
    Unknown | 9 | 4 | 13
    MISSING | 13 | 3 | 16
Prior stem cell transplant [Count of Participants; unit: Participants]
  Autologous | 114 | 57 | 171
  Allogeneic | 2 | 0 | 2
  Syngeneic | 0 | 0 | 0
  MISSING | 78 | 40 | 118

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the number of days from the date the participant was randomized to the date of the first documented progressive disease (PD) as determined by an Independent Review Committee (IRC) or death due to any cause, whichever occurs first. PFS was analyzed by Kaplan-Meier methodology.
Time Frame: Median duration of follow-up was 28.6 months for the venetoclax group and 28.6 months for the placebo group
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 194 | 97
months | 23.2 [15.3 to 27.5] | 11.5 [9.6 to 15.0]
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; Stratified Analysis; Stratification factors: Prior exposure to proteasome inhibitors (naïve versus sensitive), and number of prior lines of therapy (1 versus 2 or 3); Test type: Superiority; p = 0.012, Log Rank; Hazard Ratio (HR) = 0.656, 95% CI 2-sided [0.471 to 0.913] — Hazard ratio was estimated by Cox proportional hazards model

2. Secondary Outcome: Very Good Partial Response (VGPR) or Better Response Rate
Description: The percentage of participants with documented best overall response of Very Good Partial Response (VGPR) or better (VGPR, Complete response [CR], or Stringent complete response [sCR]) per 2016 standard International Myeloma Working Group (IMWG) criteria as determined by an Independent Review Committee (IRC) was computed.
Time Frame: Response was assessed at Cycle 1, Day 1, and on Day 1 of every cycle thereafter; median time on follow-up was 28.6 months for the venetoclax group and 28.6 months for the placebo group
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 194 | 97
percentage of participants | 60.3 [53.1 to 67.2] | 38.1 [28.5 to 48.6]
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Progression-Free Survival (PFS) in Participants With High B-cell Lymphoma 2 (BCL-2) Expression
Description: PFS is defined as the number of days from the date the participant was randomized to the date of the first documented progressive disease (PD) per investigator assessment or death due to any cause, whichever occurs first. PFS was analyzed by Kaplan-Meier methodology.
  BCL-2 expression was determined through central laboratory testing by immunohistochemistry (IHC) and based on a pre-specified scoring algorithm. High clinical score of 2+: ≥50% of tumor cells with moderate or higher cytoplasmic staining but < 50% of tumor cells with strong staining intensity; high clinical score of 3+: ≥50% of tumor cells with strong cytoplasmic staining.
Time Frame: Median duration of follow-up was 28.6 months for the venetoclax group and 28.6 months for the placebo group
Population: Intent-To-Treat (ITT) analysis set: all randomized participants, analyzed by treatment group assignment given at the time of randomization who had high BCL-2 expression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 93 | 47
months | 23.8 [19.5 to 34.7] | 11.4 [9.1 to 15.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the number of days from the participant's date of first documented response (partial response [PR] or better) to the date of first documented progressive disease (PD) as determined by an Independent Review Committee (IRC) or death due to multiple myeloma, whichever occurs first. DOR was analyzed by Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 158 | 67
months | NA [22.8 to NA] — Not estimable/calculable due to low number of participants with events | 12.8 [10.6 to 15.5]
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.508, 95% CI 2-sided [0.343 to 0.753] — Hazard ratio was estimated by Cox proportional hazards model

5. Secondary Outcome: Mean Change From Baseline in Brief Pain Inventory - Short Form (BPI-SF) Worst Pain
Description: The BPI-SF is a pain-specific measure developed to assess patient-reported severity (or intensity) of pain (4 items) and the impact of pain on daily functioning (7 items) in patients with cancer pain. The four pain severity items assess pain at its "worst in last 24 hours," "least in last 24 hours," "average," and "now" (current pain). For these items, participants are asked to rate their pain on an 11-point numeric rating scale with anchors of 0 (no pain) and 10 (pain as bad as you can imagine). The Worst Pain scores range from 0 to 10, with higher scores indicating severe pain. Negative changes from baseline indicate improvement.
Time Frame: Baseline; Cycle 3 (Cycles 1 - 8 are 21 days, Cycles 9 and beyond are 35 days) through Cycle 47, collected on Day 1 of every other cycle and at the Treatment Completion Visit (TCV) while participant is on treatment
Population: Intent-To-Treat (ITT) analysis set: all randomized participants, analyzed by treatment group assignment given at the time of randomization; participants who have both baseline and post-baseline values are included in the analysis at each visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 184 | 92
units on a scale
  Cycle 3, Day 1: number analyzed (Participants) | 162 | 79
  Cycle 3, Day 1 | -0.6 (2.59) | -0.5 (2.46)
  Cycle 5, Day 1: number analyzed (Participants) | 140 | 70
  Cycle 5, Day 1 | 0.0 (2.65) | -0.2 (3.15)
  Cycle 7, Day 1: number analyzed (Participants) | 126 | 70
  Cycle 7, Day 1 | -0.1 (2.56) | 0.2 (2.98)
  Cycle 9, Day 1: number analyzed (Participants) | 113 | 65
  Cycle 9, Day 1 | -0.2 (3.11) | 0.0 (2.88)
  Cycle 11, Day 1: number analyzed (Participants) | 98 | 55
  Cycle 11, Day 1 | -0.4 (2.57) | 0.1 (3.45)
  Cycle 13, Day 1: number analyzed (Participants) | 82 | 43
  Cycle 13, Day 1 | -0.2 (2.71) | -0.1 (3.22)
  Cycle 15, Day 1: number analyzed (Participants) | 76 | 31
  Cycle 15, Day 1 | -0.2 (2.92) | -0.0 (3.08)
  Cycle 17, Day 1: number analyzed (Participants) | 66 | 27
  Cycle 17, Day 1 | -0.3 (2.54) | -0.1 (2.06)
  Cycle 19, Day 1: number analyzed (Participants) | 67 | 22
  Cycle 19, Day 1 | -0.1 (2.59) | -0.2 (1.95)
  Cycle 21, Day 1: number analyzed (Participants) | 59 | 18
  Cycle 21, Day 1 | -0.1 (2.39) | -0.3 (2.89)
  Cycle 23, Day 1: number analyzed (Participants) | 55 | 17
  Cycle 23, Day 1 | -0.0 (3.20) | -0.2 (2.61)
  Cycle 25, Day 1: number analyzed (Participants) | 47 | 13
  Cycle 25, Day 1 | 0.4 (2.65) | 0.2 (3.00)
  Cycle 27, Day 1: number analyzed (Participants) | 37 | 14
  Cycle 27, Day 1 | 0.2 (2.53) | 0.1 (1.92)
  Cycle 29, Day 1: number analyzed (Participants) | 40 | 15
  Cycle 29, Day 1 | -0.2 (2.83) | 0.3 (2.15)
  Cycle 31, Day 1: number analyzed (Participants) | 39 | 9
  Cycle 31, Day 1 | 0.0 (3.11) | 0.6 (1.33)
  Cycle 33, Day 1: number analyzed (Participants) | 37 | 7
  Cycle 33, Day 1 | -0.2 (2.88) | 0.4 (1.40)
  Cycle 35, Day 1: number analyzed (Participants) | 34 | 6
  Cycle 35, Day 1 | 0.1 (2.77) | -0.2 (1.33)
  Cycle 37, Day 1: number analyzed (Participants) | 31 | 4
  Cycle 37, Day 1 | 0.4 (2.78) | 1.5 (2.65)
  Cycle 39, Day 1: number analyzed (Participants) | 26 | 3
  Cycle 39, Day 1 | 0.1 (2.70) | -0.3 (1.15)
  Cycle 41, Day 1: number analyzed (Participants) | 21 | 3
  Cycle 41, Day 1 | 0.1 (3.00) | 0.3 (1.15)
  Cycle 43, Day 1: number analyzed (Participants) | 17 | 2
  Cycle 43, Day 1 | -0.1 (3.07) | 0.5 (0.71)
  Cycle 45, Day 1: number analyzed (Participants) | 9 | 2
  Cycle 45, Day 1 | -0.7 (3.64) | 1.0 (0.00)
  Cycle 47, Day 1: number analyzed (Participants) | 4 | 1
  Cycle 47, Day 1 | -2.8 (3.77) | 1.0
  Final visit: number analyzed (Participants) | 175 | 87
  Final visit | 0.3 (3.28) | 0.4 (3.55)

6. Secondary Outcome: Mean Change From Baseline in Physical Functioning Scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status/quality of life scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). For the Physical Functioning scale, participants rate five items on a four-point scale, with 1 as "not at all" and 4 as "very much." The Physical Functioning Scale scores range from 0 to 100 and were calculated per the EORTC QLQ-C30 Scoring Manual (3rd edition), version 3.0. A high scale score represents high/healthy level of functioning. Positive changes from baseline indicate improvement.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 184 | 92
units on a scale
  Cycle 3, Day 1: number analyzed (Participants) | 161 | 79
  Cycle 3, Day 1 | -5.0 (18.22) | -4.6 (19.50)
  Cycle 5, Day 1: number analyzed (Participants) | 140 | 70
  Cycle 5, Day 1 | -3.9 (18.38) | -7.8 (21.50)
  Cycle 7, Day 1: number analyzed (Participants) | 126 | 70
  Cycle 7, Day 1 | -6.1 (20.19) | -8.6 (19.76)
  Cycle 9, Day 1: number analyzed (Participants) | 114 | 65
  Cycle 9, Day 1 | -3.5 (19.54) | -8.0 (20.01)
  Cycle 11, Day 1: number analyzed (Participants) | 99 | 55
  Cycle 11, Day 1 | -1.5 (15.92) | -7.5 (18.46)
  Cycle 13, Day 1: number analyzed (Participants) | 83 | 43
  Cycle 13, Day 1 | -3.2 (16.57) | -8.8 (22.85)
  Cycle 15, Day 1: number analyzed (Participants) | 77 | 31
  Cycle 15, Day 1 | -2.3 (18.72) | -7.3 (22.27)
  Cycle 17, Day 1: number analyzed (Participants) | 67 | 27
  Cycle 17, Day 1 | -1.8 (16.23) | -8.6 (19.90)
  Cycle 19, Day 1: number analyzed (Participants) | 68 | 22
  Cycle 19, Day 1 | -2.5 (19.30) | -7.0 (19.35)
  Cycle 21, Day 1: number analyzed (Participants) | 59 | 18
  Cycle 21, Day 1 | -1.5 (17.81) | -8.5 (20.43)
  Cycle 23, Day 1: number analyzed (Participants) | 55 | 17
  Cycle 23, Day 1 | -3.4 (20.32) | -7.5 (20.53)
  Cycle 25, Day 1: number analyzed (Participants) | 48 | 13
  Cycle 25, Day 1 | -3.8 (17.28) | 0.5 (23.95)
  Cycle 27, Day 1: number analyzed (Participants) | 38 | 14
  Cycle 27, Day 1 | -8.6 (21.69) | -3.3 (18.44)
  Cycle 29, Day 1: number analyzed (Participants) | 40 | 15
  Cycle 29, Day 1 | -8.7 (21.25) | -4.0 (19.81)
  Cycle 31, Day 1: number analyzed (Participants) | 40 | 9
  Cycle 31, Day 1 | -2.8 (17.98) | 2.2 (18.56)
  Cycle 33, Day 1: number analyzed (Participants) | 38 | 7
  Cycle 33, Day 1 | -4.0 (22.76) | -4.8 (23.64)
  Cycle 35, Day 1: number analyzed (Participants) | 35 | 6
  Cycle 35, Day 1 | -7.0 (16.64) | 4.4 (18.70)
  Cycle 37, Day 1: number analyzed (Participants) | 31 | 4
  Cycle 37, Day 1 | -7.5 (22.49) | 15.0 (14.78)
  Cycle 39, Day 1: number analyzed (Participants) | 27 | 3
  Cycle 39, Day 1 | -10.1 (18.80) | 8.9 (10.18)
  Cycle 41, Day 1: number analyzed (Participants) | 22 | 3
  Cycle 41, Day 1 | -13.0 (25.65) | 13.3 (23.09)
  Cycle 43, Day 1: number analyzed (Participants) | 17 | 2
  Cycle 43, Day 1 | -7.8 (23.12) | 13.3 (18.86)
  Cycle 45, Day 1: number analyzed (Participants) | 10 | 2
  Cycle 45, Day 1 | -1.3 (10.33) | 13.3 (18.86)
  Cycle 47, Day 1: number analyzed (Participants) | 4 | 1
  Cycle 47, Day 1 | 0.0 (14.40) | 0.0
  Final visit: number analyzed (Participants) | 175 | 87
  Final visit | -11.8 (22.85) | -10.0 (21.52)

7. Secondary Outcome: Mean Change From Baseline in Global Health Status/Quality of Life Scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status/quality of life scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). For the Global Health Status/Quality of Life scale, participants rate two items on a seven point scale, with 1 as "very poor" and 7 as "excellent." The Global Health Status/Quality of Life scale ranges from 0 to 100 and was calculated per the EORTC QLQ-C30 Scoring Manual (3rd edition), version 3.0. A high score for the global health status/QoL represents a high QoL. Positive changes from baseline indicate improvement.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 184 | 92
units on a scale
  Cycle 3, Day 1: number analyzed (Participants) | 161 | 79
  Cycle 3, Day 1 | -1.9 (22.75) | -2.2 (22.63)
  Cycle 5, Day 1: number analyzed (Participants) | 140 | 70
  Cycle 5, Day 1 | -5.1 (26.74) | -2.5 (23.54)
  Cycle 7, Day 1: number analyzed (Participants) | 126 | 70
  Cycle 7, Day 1 | -8.3 (26.76) | -6.7 (24.56)
  Cycle 9, Day 1: number analyzed (Participants) | 114 | 65
  Cycle 9, Day 1 | -6.9 (26.33) | -6.7 (24.22)
  Cycle 11, Day 1: number analyzed (Participants) | 99 | 55
  Cycle 11, Day 1 | -0.5 (25.58) | -5.2 (25.38)
  Cycle 13, Day 1: number analyzed (Participants) | 83 | 43
  Cycle 13, Day 1 | -1.0 (25.05) | -1.7 (22.24)
  Cycle 15, Day 1: number analyzed (Participants) | 77 | 31
  Cycle 15, Day 1 | -4.9 (26.09) | 0.5 (23.56)
  Cycle 17, Day 1: number analyzed (Participants) | 67 | 27
  Cycle 17, Day 1 | -5.1 (24.91) | -7.7 (21.55)
  Cycle 19, Day 1: number analyzed (Participants) | 68 | 22
  Cycle 19, Day 1 | -1.3 (19.51) | 0.8 (26.09)
  Cycle 21, Day 1: number analyzed (Participants) | 59 | 18
  Cycle 21, Day 1 | -6.6 (26.16) | -5.6 (20.01)
  Cycle 23, Day 1: number analyzed (Participants) | 55 | 17
  Cycle 23, Day 1 | -2.9 (23.20) | -1.0 (22.99)
  Cycle 25, Day 1: number analyzed (Participants) | 48 | 13
  Cycle 25, Day 1 | -4.7 (26.29) | -4.5 (24.68)
  Cycle 27, Day 1: number analyzed (Participants) | 38 | 14
  Cycle 27, Day 1 | -9.0 (24.46) | 4.2 (26.70)
  Cycle 29, Day 1: number analyzed (Participants) | 40 | 15
  Cycle 29, Day 1 | -6.9 (24.67) | -1.1 (26.33)
  Cycle 31, Day 1: number analyzed (Participants) | 40 | 9
  Cycle 31, Day 1 | -4.8 (26.48) | 5.6 (35.36)
  Cycle 33, Day 1: number analyzed (Participants) | 38 | 7
  Cycle 33, Day 1 | -7.7 (27.22) | -7.1 (22.79)
  Cycle 35, Day 1: number analyzed (Participants) | 35 | 6
  Cycle 35, Day 1 | -3.8 (24.03) | 4.2 (29.23)
  Cycle 37, Day 1: number analyzed (Participants) | 31 | 4
  Cycle 37, Day 1 | -13.7 (29.86) | 10.4 (12.50)
  Cycle 39, Day 1: number analyzed (Participants) | 27 | 3
  Cycle 39, Day 1 | -9.3 (28.05) | 0.0 (0.00)
  Cycle 41, Day 1: number analyzed (Participants) | 22 | 3
  Cycle 41, Day 1 | -11.0 (30.47) | 8.3 (8.33)
  Cycle 43, Day 1: number analyzed (Participants) | 17 | 2
  Cycle 43, Day 1 | 2.0 (28.95) | -8.3 (23.57)
  Cycle 45, Day 1: number analyzed (Participants) | 10 | 2
  Cycle 45, Day 1 | -1.7 (33.75) | 4.2 (5.89)
  Cycle 47, Day 1: number analyzed (Participants) | 4 | 1
  Cycle 47, Day 1 | 10.4 (22.95) | -8.3
  Final visit: number analyzed (Participants) | 175 | 87
  Final visit | -8.1 (26.40) | -6.7 (28.50)

8. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcomes Measurement Information System [PROMIS] Cancer Fatigue Short Form [SF] Score
Description: PROMIS Cancer Fatigue SF is a seven item questionnaire that assesses the impact and experience of fatigue over the past 7 days. All questions employ the following five response options: 1 = Not at all, 2 = A little bit, 3 = Somewhat, 4 = Quite a bit, and 5 = Very much. The total raw score is the sum of the responses to each question and is converted to a T-score. The T-score re-scales the total raw score to a standardized score with a mean of 50 and a standard deviation of 10. The [PROMIS] Cancer Fatigue Short Form [SF] 7a T-Scores range from 29.4 to 83.2, with higher scores indicating more fatigue. Negative changes from baseline indicate improvement.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 185 | 92
T-score
  Cycle 3, Day 1: number analyzed (Participants) | 163 | 79
  Cycle 3, Day 1 | 2.2 (9.54) | 1.8 (8.12)
  Cycle 5, Day 1: number analyzed (Participants) | 141 | 70
  Cycle 5, Day 1 | 3.3 (9.25) | 2.4 (10.34)
  Cycle 7, Day 1: number analyzed (Participants) | 126 | 70
  Cycle 7, Day 1 | 3.2 (9.28) | 2.6 (9.70)
  Cycle 9, Day 1: number analyzed (Participants) | 114 | 65
  Cycle 9, Day 1 | 2.3 (8.90) | 2.6 (8.67)
  Cycle 11, Day 1: number analyzed (Participants) | 99 | 55
  Cycle 11, Day 1 | 0.6 (8.54) | 3.1 (8.98)
  Cycle 13, Day 1: number analyzed (Participants) | 83 | 43
  Cycle 13, Day 1 | 1.8 (8.03) | 2.3 (6.97)
  Cycle 15, Day 1: number analyzed (Participants) | 77 | 31
  Cycle 15, Day 1 | 1.5 (8.84) | 2.1 (7.66)
  Cycle 17, Day 1: number analyzed (Participants) | 67 | 27
  Cycle 17, Day 1 | 1.2 (8.11) | 2.6 (8.05)
  Cycle 19, Day 1: number analyzed (Participants) | 68 | 22
  Cycle 19, Day 1 | 0.7 (8.52) | 0.9 (9.32)
  Cycle 21, Day 1: number analyzed (Participants) | 59 | 18
  Cycle 21, Day 1 | 1.6 (8.58) | 1.2 (7.66)
  Cycle 23, Day 1: number analyzed (Participants) | 55 | 17
  Cycle 23, Day 1 | 2.0 (8.08) | 1.5 (8.83)
  Cycle 25, Day 1: number analyzed (Participants) | 48 | 13
  Cycle 25, Day 1 | 2.0 (8.59) | -0.1 (8.73)
  Cycle 27, Day 1: number analyzed (Participants) | 38 | 14
  Cycle 27, Day 1 | 3.4 (8.19) | -0.1 (9.59)
  Cycle 29, Day 1: number analyzed (Participants) | 40 | 15
  Cycle 29, Day 1 | 3.9 (8.07) | 0.8 (8.51)
  Cycle 31, Day 1: number analyzed (Participants) | 40 | 9
  Cycle 31, Day 1 | 2.8 (8.43) | -0.3 (9.15)
  Cycle 33, Day 1: number analyzed (Participants) | 38 | 7
  Cycle 33, Day 1 | 2.0 (8.93) | 3.7 (9.17)
  Cycle 35, Day 1: number analyzed (Participants) | 35 | 6
  Cycle 35, Day 1 | 3.4 (9.27) | 1.1 (7.22)
  Cycle 37, Day 1: number analyzed (Participants) | 31 | 4
  Cycle 37, Day 1 | 4.1 (9.72) | -3.0 (11.72)
  Cycle 39, Day 1: number analyzed (Participants) | 27 | 3
  Cycle 39, Day 1 | 3.6 (8.12) | 4.1 (2.82)
  Cycle 41, Day 1: number analyzed (Participants) | 22 | 3
  Cycle 41, Day 1 | 3.3 (8.69) | -0.7 (6.90)
  Cycle 43, Day 1: number analyzed (Participants) | 17 | 2
  Cycle 43, Day 1 | 5.3 (9.28) | 4.4 (1.91)
  Cycle 45, Day 1: number analyzed (Participants) | 10 | 2
  Cycle 45, Day 1 | -0.3 (7.99) | 1.8 (0.28)
  Cycle 47, Day 1: number analyzed (Participants) | 4 | 1
  Cycle 47, Day 1 | -2.5 (6.30) | 0.0
  Final visit: number analyzed (Participants) | 176 | 87
  Final visit | 5.0 (10.95) | 2.9 (9.96)

9. Secondary Outcome: Overall Survival (OS).
Description: OS is defined as the number of days from the date of randomization to the date of death due to any cause. All events of death were to be included, regardless of whether the event occurred while the participant was still taking study drug or after the participant discontinued study drug. If a participant is not known to have died, OS was censored at the date of last contact. The distribution of OS was estimated using Kaplan-Meier methodology.
Time Frame: Median duration of follow-up was 45.6 months for the venetoclax group and 45.6 months for the placebo group
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 194 | 97
months | NA [44.4 to NA] — Not estimable/calculable due to low number of participants with events | NA [44.0 to NA] — Not estimable/calculable due to low number of participants with events
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.385, Log Rank; Hazard Ratio (HR) = 1.191, 95% CI 2-sided [0.802 to 1.770] — Hazard ratio was estimated by Cox proportional hazards model

10. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days from the date of randomization to the date of first documented progressive disease (PD) as determined by an Independent Review Committee (IRC) or death due to multiple myeloma, whichever occurs first. TTP was analyzed by Kaplan-Meier methodology.
Time Frame: Median time on follow-up up was 28.6 months for the venetoclax group and 28.6 months for the placebo group
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 194 | 97
months | 25.4 [20.6 to NA] — Not estimable/calculable due to low number of participants with events | 12.2 [9.9 to 15.0]
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.571, 95% CI 2-sided [0.405 to 0.805] — Hazard ratio was estimated by Cox proportional hazards model

11. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as the percentage of participants with documented best overall response of Partial Response (PR) or better (PR, Very good partial response [VGPR], Complete response [CR], or Stringent complete response [sCR]) per International Myeloma Working Group (IMWG) criteria as determined by an Independent Review Committee (IRC).
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 194 | 97
percentage of participants | 81.4 [75.2 to 86.7] | 69.1 [58.9 to 78.1]
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel

12. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate is defined as the percentage of participants who have negative MRD by bone marrow aspirate at any time point after randomization and before progression or starting subsequent therapy. MRD negativity was defined at 10^-5 threshold (less than one residual myeloma cell per 10^5 total nucleated cells) as measured by centralized testing of bone marrow aspirate by Next Generation Sequencing (NGS). MRD positive participants include those of which all tested samples were found to be MRD positive or indeterminate. Participants with missing or unevaluable MRD status were considered as MRD positive.
Time Frame: Assessed at Screening; to confirm a stringent Complete Response (sCR) or Complete Response (CR); at 6 months and 12 months post-confirmed CR/sCR
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
Number analyzed (Participants) | 194 | 97
percentage of participants | 15.5 [10.7 to 21.3] | 2.1 [0.3 to 7.3]
Statistical Analysis 1: Comparison: Venetoclax + Bortezomib and Dexamethasone vs Placebo + Bortezomib and Dexamethasone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow-up was 48.4 months for the venetoclax group and 47.2 months for the placebo group. TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean time on venetoclax was 582.2 days and mean time on placebo was 431.3 days.
Description: All-cause mortality is reported for all enrolled participants; one participant in each group did not receive treatment.
Arm/Group | Venetoclax + Bortezomib and Dexamethasone | Placebo + Bortezomib and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 81/194 | 36/97
Serious Adverse Events (participants affected / at risk) | 115/193 | 53/96
Other Adverse Events (participants affected / at risk) | 191/193 | 95/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Bortezomib and Dexamethasone (N=193) | Placebo + Bortezomib and Dexamethasone (N=96)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 4 (6) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 2 (2) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
TOXIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 3 (3) | 3 (4)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 2 (2)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (5) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 2 (2) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 (2) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
BILIARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 6 (9) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS B REACTIVATION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 3 (3) | 0 (0)
INFECTION (Infections and infestations) | 2 (2) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (2)
INFLUENZA (Infections and infestations) | 3 (3) | 4 (4)
LARGE INTESTINE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LISTERIOSIS (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (9) | 5 (7)
MEDICAL DEVICE SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NECROTISING FASCIITIS (Infections and infestations) | 1 (2) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PERIODONTITIS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 35 (53) | 14 (19)
PNEUMONIA ADENOVIRAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA INFLUENZAL (Infections and infestations) | 4 (4) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 6 (8) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (2) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (2) | 0 (0)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
BONE LESION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
SACRAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
VERTEBRAL WEDGING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MEDIASTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AUTONOMIC NEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
EMBOLIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 4 (4) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 3 (4)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (3) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 5 (5) | 2 (2)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Bortezomib and Dexamethasone (N=193) | Placebo + Bortezomib and Dexamethasone (N=96)
ANAEMIA (Blood and lymphatic system disorders) | 48 (73) | 23 (31)
LYMPHOPENIA (Blood and lymphatic system disorders) | 19 (54) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 54 (183) | 9 (16)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 53 (120) | 34 (78)
PALPITATIONS (Cardiac disorders) | 5 (6) | 6 (6)
CATARACT (Eye disorders) | 24 (33) | 11 (17)
VISION BLURRED (Eye disorders) | 8 (9) | 5 (5)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 10 (12) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 15 (17) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 23 (38) | 8 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 20 (26) | 7 (9)
CONSTIPATION (Gastrointestinal disorders) | 68 (89) | 29 (35)
DIARRHOEA (Gastrointestinal disorders) | 114 (282) | 46 (79)
DYSPEPSIA (Gastrointestinal disorders) | 24 (28) | 9 (10)
FLATULENCE (Gastrointestinal disorders) | 12 (13) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 10 (16) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 73 (112) | 22 (28)
STOMATITIS (Gastrointestinal disorders) | 8 (9) | 5 (5)
VOMITING (Gastrointestinal disorders) | 38 (62) | 17 (27)
ASTHENIA (General disorders) | 30 (39) | 2 (2)
FATIGUE (General disorders) | 63 (90) | 31 (43)
INFLUENZA LIKE ILLNESS (General disorders) | 10 (20) | 7 (10)
INJECTION SITE REACTION (General disorders) | 5 (6) | 5 (5)
MALAISE (General disorders) | 10 (10) | 2 (3)
OEDEMA PERIPHERAL (General disorders) | 38 (57) | 20 (25)
PAIN (General disorders) | 4 (4) | 5 (5)
PYREXIA (General disorders) | 31 (40) | 11 (13)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 11 (13) | 0 (0)
BRONCHITIS (Infections and infestations) | 30 (45) | 15 (20)
CONJUNCTIVITIS (Infections and infestations) | 22 (26) | 7 (8)
INFLUENZA (Infections and infestations) | 28 (38) | 4 (11)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 (19) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 35 (92) | 8 (15)
PNEUMONIA (Infections and infestations) | 14 (18) | 3 (3)
SINUSITIS (Infections and infestations) | 10 (14) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 55 (149) | 25 (46)
URINARY TRACT INFECTION (Infections and infestations) | 15 (16) | 4 (4)
CONTUSION (Injury, poisoning and procedural complications) | 12 (13) | 6 (7)
FALL (Injury, poisoning and procedural complications) | 22 (25) | 8 (11)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 15 (22) | 9 (13)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 17 (23) | 5 (7)
BLOOD CREATININE INCREASED (Investigations) | 14 (18) | 2 (5)
C-REACTIVE PROTEIN INCREASED (Investigations) | 13 (15) | 3 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 21 (54) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 33 (78) | 15 (50)
WEIGHT DECREASED (Investigations) | 11 (15) | 2 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 42 (60) | 13 (14)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 20 (29) | 8 (12)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 16 (21) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 32 (49) | 8 (12)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 12 (14) | 4 (11)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 (37) | 12 (13)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 43 (48) | 17 (23)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 15 (20) | 5 (5)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 17 (22) | 8 (8)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 17 (19) | 10 (10)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 9 (12) | 6 (6)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 13 (13) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 25 (32) | 14 (15)
DIZZINESS (Nervous system disorders) | 34 (44) | 10 (11)
DYSGEUSIA (Nervous system disorders) | 16 (18) | 5 (5)
HEADACHE (Nervous system disorders) | 31 (50) | 16 (19)
HYPOAESTHESIA (Nervous system disorders) | 14 (16) | 8 (12)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 59 (84) | 27 (35)
PARAESTHESIA (Nervous system disorders) | 18 (24) | 5 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 36 (60) | 24 (36)
INSOMNIA (Psychiatric disorders) | 56 (73) | 29 (33)
COUGH (Respiratory, thoracic and mediastinal disorders) | 44 (65) | 20 (27)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 22 (33) | 15 (21)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (8)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (10)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 5 (8)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (25) | 4 (5)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 33 (47) | 8 (11)
RASH (Skin and subcutaneous tissue disorders) | 25 (27) | 4 (5)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
HYPERTENSION (Vascular disorders) | 20 (23) | 15 (18)
HYPOTENSION (Vascular disorders) | 23 (25) | 4 (5)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 13 (15) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02755597/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02755597/SAP_001.pdf